CLINICAL TRIAL: NCT01873079
Title: Prevention of Delayed Post-sphincterotomy Bleeding by High Dose Proton Pump Inhibitor
Brief Title: PPI for Prevention of Post-sphincterotomy Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEUNG Wai Keung, Clinical Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ERCP-PPI ver. 2
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Bleeding; ERCP
Keywords: ERCP; sphincterotomy; proton pump inhibitor
MeSH Terms: conditions — Hemorrhage | interventions — Esomeprazole; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esomeprazole (Active Comparator): esomeprazole 40mg bd for 10 days
  Interventions: Drug: Esomeprazole
- Standard care (Sham Comparator): No other study drug or placebo will be given
  Interventions: Other: Standard care

INTERVENTIONS:
Drug: Esomeprazole
  Other Names: Nexium
  Arms: Esomeprazole
Other: Standard care — No PPI or other study medication given
  Arms: Standard care

SUMMARY:
Endoscopic biliary sphincterotomy is a common and important procedure for biliary access and therapy during endoscopic retrograde cholangiopancreatography (ERCP). Bleeding is one of the important complications related to sphincterotomy. This study determines the role of proton pump inhibitor (PPI) in preventing post-sphincterotomy bleeding in patients undergoing ERCP and sphincterotomy.

DETAILED DESCRIPTION:
Eligible patients will be randomized to receive either high dose PPI or standard care. PPI will be given before ERCP and continue for one week after the sphincterotomy.

Both overt and occult bleeding will be documented up to 10 days after the sphincterotomy. Bleeding rates of the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing ERCP who will require sphincterotomy

Exclusion Criteria:

* Previous sphincterotomy/papillotomy
* Previous Polya gastrectomy
* Patients on maintenance PPI
* Pregnant and lactating women
* Age <18 years
* Previous liver transplant
* unable to consent for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2013-04; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with bleeding after sphincterotomy | 10 days

SECONDARY OUTCOMES:
Proportion of patients who require transfusion, endoscopic hemostasis and other intervention to control bleeding | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Wai K Leung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China